CLINICAL TRIAL: NCT07303010
Title: The Effect of Cryotherapy on Treatment Outcomes for Pulpotomy in Permanent Mature Carious Posterior Teeth: A Randomized Controlled Trial
Brief Title: The Effect of Cryotherapy on Treatment Outcomes for Pulpotomy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sirawut Hiran-us (Other)
Responsible Party: Sponsor-Investigator, Sirawut Hiran-us, Associate Orofessor, Chulalongkorn University
Organization: Chulalongkorn University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BBC 33/2025
Record Dates: First submitted 2025-12-06; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Carious Teeth
Keywords: pulpotomy; cryotherapy
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Addition of Cryotherapy on pulpotomy (Experimental): Experimental: Addition of Cryotherapy on pulpotomy After hemostasis is achieved, the pulpotomy area is irrigated for 5 minutes with normal saline solution, which is kept in the refrigerator set to 2.5°C (measuring with thermometer and record) by using a disposable insulated 5 ml syringe and 21-gauge needle is placed 1-2 mm above the root canal orifices and is constantly moved in a circular motion: 5 ml in each of 4 syringes, administered every 1.25 minutes per syringe.
  Interventions: Other: Addition of Cryotherapy on pulpotomy
- Rountine pulpotomy (No Intervention): No Intervention: Rountine pulpotomy

INTERVENTIONS:
Other: Addition of Cryotherapy on pulpotomy — Experimental: Addition of Cryotherapy on pulpotomy After hemostasis is achieved, the pulpotomy area is irrigated for 5 minutes with normal saline solution, which is kept in the refrigerator set to 2.5°C (measuring with thermometer and record) by using a disposable insulated 5 ml syringe and 21-gauge needle is placed 1-2 mm above the root canal orifices and is constantly moved in a circular motion: 5 ml in each of 4 syringes, administered every 1.25 minutes per syringe.
  Arms: Addition of Cryotherapy on pulpotomy

SUMMARY:
The goal of this clinical trial is to investigate the effect of cryotherapy on treatment outcome for pulpotomny in permanent mature carious posterior teeth. The main question is: Do cryotherapy improve treatment outcome in interested samples?

[primary hypothesis or outcome measure 1] Treatment outcome by clinical and radiographic examination.

Treatment outcome from different groups will be compared at designated time points.

DETAILED DESCRIPTION:
Materials and methods Study design and setting This study is a prospective, single-center, double-blinded, parallel-group, randomized controlled trial conducted at the Dental Department, Yala Hospital. All clinical procedures are performed by a single trained operator. Clinical outcome evaluations are carried out by the same operator, while radiographic outcome evaluations are conducted by an experienced endodontist. To maintain blinding during periapical evaluation, the crown of each tooth is masked.

Study participants Inclusion Criteria

* Healthy patients aged at least 18 years old with deep or extremely deep carious lesions in mature permanent posterior teeth diagnose with asymptomatic or symptomatic irreversible pulpitis. Diagnoses are confirmed using Electric Pulp Test(EPT) and cold test. Pulpal and periapical diagnoses are based on terminology from the American Association of Endodontists (AAE, 2013).
* Teeth are restorable with direct composite restoration. Exclusion Criteria
* Teeth with subgingival caries and/or clinical attachment loss more than 3 mm and probing depth more than 4 mm.
* Negative responses to pulp sensibility tests, presence of sinus tracts, swelling, non-restorable crowns, immature roots, or no pulp exposure following complete caries removal in case of pre-operative diagnosis as asymptomatic irreversible pulpitis.
* Patients with systemic diseases involving bleeding disorders such as hemophilia, Von Willebrand disease, platelet disorders. And patients under taking all kind of anticoagulant and anti-platelet.
* Known allergies to non-steroidal anti-inflammatory drugs (NSAIDs).
* Pregnant or lactating patients.
* Teeth with pulpal obliteration.
* Necrotic pulp is found after access opening.
* Bleed cannot be stopped within 8 minutes after full pulpotomy26,27 Treatment procedure A comprehensive medical and dental history is taken before treatment. Preoperative data, including age, sex and tooth number are recorded in a predesigned patient's chart. The treatment, the study design, alternative treatment modalities, potential benefits, risks, and follow-up protocol are explained to the qualifying patients and informed consent is obtained from the voluntary patients who are willing to participate in the study.

Sample size calculation The sample size was calculated based on a suspected difference of 25% in the success rate between the control and cryotherapy group in inferior alveolar nerve block35 using n4Studies with a 80% power, a 5% α error. The minimum sample size was calculated to be 122. Considering patients lost to follow-up, a total of 140 teeth from different patients are included in this study.

Randomization and masking Block randomization with variable 4 block sizes is used to generate a sequence of random numbers for allocating the patients equally into two study groups. Each random blocks are sealed in an opaque envelope which is opened at the beginning of the clinical trial by dental assistant who the one only know the intervention and prepare the intervention for operator. New block will be open after all the patient in the previous block was completed and repeat until the end of the clinical trials to ensure the equality of group distribution: The VTP with and without cryotherapy intervention groups.

Intervention

All the treatment is carried out by a single operator under magnification(3x loupes) and illumination. All the patients received a topical anesthesia before local anesthesia. An inferior alveolar nerve block (1.8 ml 2% Lidocaine with epinephrine 1:100,000) + buccal infiltration (1.7 ml 4% Articaine with epinephrine 1:100,000) for mandibular teeth, buccal infiltration (1.8 ml 2% Lidocaine with epinephrine 1:100,000) for maxillary teeth. The anesthesia is confirmed by negative response to EPT. The pulpotomy procedure is performed under rubber dam isolation in a single visit. If the patient experienced pain during the procedure, an additional anesthesia is used to achieve profound pulpal anesthesia by intraligament injection with 0.3 ml 2% Lidocaine with epinephrine 1:100,000. The operating field is disinfected with iodine and alcohol. A cylindrical diamond airotor operates under air water coolant to outline the cavity. Low speed round steel bur and a spoon excavator are used to remove the soft carious dentine using nonselective caries removal from the periphery towards the centre of the carious lesion. The deepest layer of carious dentine is thereafter disinfected with 2 ml of 2.5% NaOCl prior to pulpal exposure. The new high-speed sterile diamond airotor is used to completely remove the coronal pulp tissue. Then rinse with of 2.5% NaOCl solution up to 8 minutes to arrest the bleeding. The time to achieve hemostasis is recorded in minutes and seconds. The diagnosis of vital inflamed pulp is confirmed by the presence of bleeding in the pulp chamber. The dental assistant will bring an insulated syringe containing different intervention as follow:

Group I (Cryotherapy): After hemostasis is achieved, the pulpotomy area is irrigated for 5 minutes with normal saline solution, which is kept in the refrigerator set to 2.5°C (measuring with thermometer) by using a disposable insulated 5 ml syringe and 21-gauge needle is placed 1-2 mm above the root canal orifices and is constantly moved in a circular motion: 5 ml in each of 4 syringes, administered every 1.25 minutes per syringe.

Group II (Control): After hemostasis is achieved, the pulpotomy area is irrigated for 5 minutes with normal saline solution, which is kept in the room temperature 25°C (measuring with thermometer) by using a disposable insulated 5 ml syringe and 21-gauge needle is placed 1-2 mm above the root canal orifices and is constantly moved in a circular motion.

In both study groups, 2 mm calcium silicate cement putty type (TFRRM) is placed as a capping agent over the residual pulp. The tooth is restored with Resin Modified Glass Ionomer Cement (RMGIC) base (Vitrebond, 3M) and composite restoration (Z350XT, 3M) and polishing in the same visit.

The full pulpotomy cases where bleeding from residual pulp cannot be arrested within 8 minutes, are excluded from the study, and pulpectomy are performed. Immediate post-operative periapical radiograph is taken.

Outcome assessment All the teeth are assessed clinically at 6 months and every year and radiographs are taken. Clinically asymptomatic teeth without any radiographic evidence of periapical rarefaction or root resorption are categorized as success in strict criteria and categorized as survival in loose criteria when clinically asymptomatic teeth with periapical rarefaction14.

Recall Clinical evaluation and periapical radiograph will be taken. The quality of the coronal restoration is checked, and the restorations are repaired if deemed necessary. In case of failed cased, the cause of failure will be identified and recorded. Proper treatment will be proposed for specific problem.

All clinical evaluation will be evaluated by the same operator who is blinded from the intervention. Clinical evaluation included

* Coronal restoration
* EPT
* Percussion
* Palpation
* Mobility
* Probing depth
* Occlusion Radiographic evaluation included
* Periapical radiograph The same operator will judge the quality of the recall radiograph which include
* 3x3 mm area covered the periapical area
* No distortion or blurred
* The image is able to interpret the periapical tissue

The blinded experienced endodontist will be evaluate the radiographic success of recall radiograph by recording as:

* Normal periapical tissue
* Thickening PDL space
* Periapical lesion

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients aged at least 18 years old with deep or extremely deep carious lesions in mature permanent posterior teeth diagnose with asymptomatic or symptomatic irreversible pulpitis. Diagnoses are confirmed using Electric Pulp Test(EPT) and cold test. Pulpal and periapical diagnoses are based on terminology from the American Association of Endodontists (AAE, 2013).
* Teeth are restorable with direct composite restoration.

Exclusion Criteria:

* Teeth with subgingival caries and/or clinical attachment loss more than 3 mm and probing depth more than 4 mm.
* Negative responses to pulp sensibility tests, presence of sinus tracts, swelling, non-restorable crowns, immature roots, or no pulp exposure following complete caries removal in case of pre-operative diagnosis as asymptomatic irreversible pulpitis.
* Patients with systemic diseases involving bleeding disorders such as hemophilia, Von Willebrand disease, platelet disorders. And patients under taking all kind of anticoagulant and anti-platelet.
* Known allergies to non-steroidal anti-inflammatory drugs (NSAIDs).
* Pregnant or lactating patients.
* Teeth with pulpal obliteration.
* Necrotic pulp is found after access opening.
* Bleed cannot be stopped within 8 minutes after full pulpotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2035-12-30 (Estimated); Study Completion 2035-12-30 (Estimated)

PRIMARY OUTCOMES:
Treatment outcome of pulpotomy | The outcomes will be evaluated as healed, healing or disease at one year after completion of treatment and annually thereafter for up to ten years, or until the patient is no longer available for follow-up.
  Determine the treatment outcome in to success or failure
  Success: No clinical sign and symptom and no abnormality of periapical tissue from radiograph
  Failure: Presence of any clinical sign or symptom or abnormality of periapical tissue from radiograph

CONTACTS AND LOCATIONS:
Overall Officials: Sirawut Hiran-us, DDS, MSc, High Grad Dip, FRCDS, Study Director — Faculty of Dentistry, Chulalongkorn University; Sawat Pojlerdarun, DDS, Higher Grad Dip, FRCDS, Principal Investigator — Yala Hospital
Locations (1):
- Yala Hospital, Yala, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Taha NA, Albakri SW. Outcome and Prognostic Factors for Partial and Full Pulpotomy in the Management of Spontaneous Symptomatic Pulpitis in Carious Mature Permanent Teeth: A Randomized Clinical Trial. J Endod. 2024 Jul;50(7):889-898. doi: 10.1016/j.joen.2024.03.012. Epub 2024 Apr 5. PMID 38583758